CLINICAL TRIAL: NCT06846450
Title: Phase 3 Trial Comparing IMRT or IMPT Plus CIRT for Patients With NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lin Kong, MD (Other)
Responsible Party: Sponsor-Investigator, Lin Kong, MD, Chief physician, Shanghai Proton and Heavy Ion Center
Organization: Shanghai Proton and Heavy Ion Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2024-70
Record Dates: First submitted 2025-02-17; First posted 2025-02-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: Proton; Photon; Carbon ion; Phase 3 Trial; Locally Advanced NPC
MeSH Terms: interventions — Induction Chemotherapy

STUDY DESIGN:
Intervention Model Description: This study adopts a web-based central randomization system. The randomization method uses minimization, with two balancing factors:
  Stage (AJCC Staging System, 9th edition): Stage I vs. Stages II/III; Response to induction chemotherapy: No induction chemotherapy vs. sensitive (CR + PR) vs. resistant (SD + PD).
  Eligible patients will be randomized in a 1:1 ratio into either the experimental group or the control group. This is an open-label study, meaning both patients and investigators are aware of the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Radiation: Intensity-modulated proton radiation therapy; Radiation: Intensity-modulated carbon ion radiation therapy; Drug: Concurrent chemotherapy; Drug: Induction chemotherapy
- Arm 2 (Active Comparator)
  Interventions: Radiation: Intensity-modulated photon radiation therapy; Radiation: Intensity-modulated carbon ion radiation therapy; Drug: Concurrent chemotherapy; Drug: Induction chemotherapy

INTERVENTIONS:
Radiation: Intensity-modulated proton radiation therapy — Intensity-modulated proton therapy, will be delivered to the high risk area with a dose of 56 GyRBE in 28 fractions, and if applicable, to the low risk area with a dose of 50.4 GyRBE in 28 fractions.
  Other Names: IMPT
  Arms: Arm 1
Radiation: Intensity-modulated photon radiation therapy — Intensity-modulated photon therapy, will be delivered to the high risk area with a dose of 56 Gy in 28 fractions, and if applicable, to the low risk area with a dose of 50.4 Gy in 28 fractions.
  Other Names: IMRT
  Arms: Arm 2
Radiation: Intensity-modulated carbon ion radiation therapy — Intensity-modulated carbon ion radiation therapy will be delivered as a boost with a dose of 17.5 GyRBE in 5 fractions to gross tumor.
  Other Names: IMCT
Drug: Concurrent chemotherapy — Concurrent chemotherapy will be administered on a weekly basis.
Drug: Induction chemotherapy — Cisplatin-based induction chemotherapy will be administered every three weekly.

SUMMARY:
The goal of this phase 3 non-inferiority trial is to compare the efficacy and toxicity of proton or photon radiation therapy plus carbon ion radiation therapy for newly diagnosed nasopharyngeal carcinoma. The main question it aims to answer is that if proton radiation therapy plus carbon ion radiation therapy is non-inferior to photon radiation therapy plus carbon ion radiation therapy in terms of therapeutic efficacy. Participants will be randomized to receive either proton radiation therapy (arm 1) or photon radiation therapy (arm 2), in addition to carbon ion radiation therapy (for both arms).

DETAILED DESCRIPTION:
This is a phase 3 randomized non-inferiority trial. The primary objective of the trial is to compare progression-free survival between proton plus carbon ion radiation therapy (arm 1) and photon plus carbon ion radiation therapy (arm 2) for patients with newly diagnosed nasopharyngeal carcinoma (NPC). The secondary objectives includes overall survival, locoregional progression-free survival, distant metastasis-free survival, physician-graded toxicities according to the CTCAE, and patients-reported outcomes. This study adopts a web-based central randomization system. The randomization method uses minimization, with two balancing factors: Stage (AJCC Staging System, 9th edition): Stage I vs. Stages II/III; Response to induction chemotherapy: No induction chemotherapy vs. sensitive (CR + PR) vs. resistant (SD + PD). Eligible patients will be randomized in a 1:1 ratio into either the experimental group or the control group. This is an open-label study, meaning both patients and investigators are aware of the treatment allocation.

Participants randomized to arm 1 will receive proton therapy with a dose of 56 GyRBE in 28 fractions, in addition to a boost delivered using carbon ion radiation therapy with a dose of 17.5 GyRBE in 5 fractions. Participants randomized to arm 2 will receive photon therapy with a dose of 56 Gy in 28 fractions, plus carbon ion radiation therapy with a dose of 17.5 GyRBE in 5 fractions. The treatment response will be evaluated according to the RECIST criteria.

Induction chemotherapy and concurrent chemotherapy will be prescribed according to disease stage.

ELIGIBILITY:
Inclusion criteria:

* Willingness to sign the written informed consent.
* Pathologically confirmed Nasopharyngeal carcinoma.
* Patients with any stage of disease except distant metastasis.
* Age: ≥ 18 and ≤ 70 years old.
* Eastern Cooperative Oncology Group score: 0-1.
* Adequate laboratory test results.
* Willingness to accept adequate contraception.

Exclusion criteria:

* Presence of distant metastasis.
* Previous radiotherapy to head and neck region.
* Previous surgery (except for biopsy) for the primary lesion or cervical lymph nodes.
* History of malignant tumor within the past 5 years.
* Presence of multiple primary tumors.
* Presence of diseases that may interfere with the evaluation of study endpoints.
* Presence of severe major organ dysfunction.
* Mental illness that may affect the understanding of informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival (PFS) defined as the time interval from randomization to death or disease progression whichever comes first.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival (OS) is defined as the time interval from randomization to death.
Locoregional progression-free survival | 3 years
  Locoregional progression-free survival (LRPFS) is defined as the time interval from randomization to death or locoregional failure whichever comes first.
Distant metastasis-free survival | 3 years
  Distant metastasis-free survival (DMFS) is defined as the time interval from randomization to death or distant metastasis whichever comes first.
Prevalence of grade ≥2 acute toxicities | 3 years
  Prevalence of grade ≥2 acute toxicities graded by CTCAE v5.
Prevalence of grade ≥3 acute toxicities | 3 years
  Prevalence of grade ≥3 acute toxicities graded by CTCAE v5.
Prevalence of grade ≥2 late toxicities | 3 years
  Prevalence of grade ≥2 late toxicities graded by CTCAE v5.
Prevalence of grade ≥3 late toxicities | 3 years
  Prevalence of grade ≥3 late toxicities graded by CTCAE v5.
Functional Assessment of Cancer Therapy | 3 years
  Patient-reported outcome, Functional Assessment of Cancer Therapy (FACT).
Xerostomia Questionnaire | 3 years
  Patient-reported outcome, Xerostomia Questionnaire (XQ).
MD Anderson Dysphagia Inventory | 3 years
  Patient-reported outcome, MD Anderson Dysphagia Inventory (MADI).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant-level data will be shared, including detailed baseline characteristics, treatment information, and follow-up data on efficacy and toxicity profile.
Supporting Information: Study Protocol, SAP
Time Frame: Anonymized IPD will be shared within 3 years after publication of the primary, secondary and safety results of the study.
Access Criteria: Data may be shared with qualified researchers who are interested in examining the efficacy and toxicity of nasopharyngeal carcinoma patients treated with particle beam radiotherapy. Pooled analysis comparing IMRT and particle beam radiotherapy will be of particular interest. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.

REFERENCES:
- [Background] Hu J, Huang Q, Gao J, Hu W, Yang J, Guan X, Qiu X, Zhang W, Kong L, Lu JJ. Mixed Photon and Carbon-Ion Beam Radiotherapy in the Management of Non-Metastatic Nasopharyngeal Carcinoma. Front Oncol. 2021 Jul 23;11:653050. doi: 10.3389/fonc.2021.653050. eCollection 2021. PMID 34367954
- [Background] Li X, Kitpanit S, Lee A, Mah D, Sine K, Sherman EJ, Dunn LA, Michel LS, Fetten J, Zakeri K, Yu Y, Chen L, Kang JJ, Gelblum DY, McBride SM, Tsai CJ, Riaz N, Lee NY. Toxicity Profiles and Survival Outcomes Among Patients With Nonmetastatic Nasopharyngeal Carcinoma Treated With Intensity-Modulated Proton Therapy vs Intensity-Modulated Radiation Therapy. JAMA Netw Open. 2021 Jun 1;4(6):e2113205. doi: 10.1001/jamanetworkopen.2021.13205. PMID 34143193
- [Background] Lewis GD, Holliday EB, Kocak-Uzel E, Hernandez M, Garden AS, Rosenthal DI, Frank SJ. Intensity-modulated proton therapy for nasopharyngeal carcinoma: Decreased radiation dose to normal structures and encouraging clinical outcomes. Head Neck. 2016 Apr;38 Suppl 1:E1886-95. doi: 10.1002/hed.24341. Epub 2015 Dec 26. PMID 26705956
- [Background] Vai A, Molinelli S, Rossi E, Iacovelli NA, Magro G, Cavallo A, Pignoli E, Rancati T, Mirandola A, Russo S, Ingargiola R, Vischioni B, Bonora M, Ronchi S, Ciocca M, Orlandi E. Proton Radiation Therapy for Nasopharyngeal Cancer Patients: Dosimetric and NTCP Evaluation Supporting Clinical Decision. Cancers (Basel). 2022 Feb 22;14(5):1109. doi: 10.3390/cancers14051109. PMID 35267415
- [Background] Minatogawa H, Yasuda K, Dekura Y, Takao S, Matsuura T, Yoshimura T, Suzuki R, Yokota I, Fujima N, Onimaru R, Shimizu S, Aoyama H, Shirato H. Potential benefits of adaptive intensity-modulated proton therapy in nasopharyngeal carcinomas. J Appl Clin Med Phys. 2021 Jan;22(1):174-183. doi: 10.1002/acm2.13128. Epub 2020 Dec 18. PMID 33338323
- [Background] Lin YH, Cheng JY, Huang BS, Luo SD, Lin WC, Chou SY, Juang PJ, Li SH, Huang EY, Wang YM. Significant Reduction in Vertebral Artery Dose by Intensity Modulated Proton Therapy: A Pilot Study for Nasopharyngeal Carcinoma. J Pers Med. 2021 Aug 22;11(8):822. doi: 10.3390/jpm11080822. PMID 34442466
- [Background] Taheri-Kadkhoda Z, Bjork-Eriksson T, Nill S, Wilkens JJ, Oelfke U, Johansson KA, Huber PE, Munter MW. Intensity-modulated radiotherapy of nasopharyngeal carcinoma: a comparative treatment planning study of photons and protons. Radiat Oncol. 2008 Jan 24;3:4. doi: 10.1186/1748-717X-3-4. PMID 18218078
- [Background] Widesott L, Pierelli A, Fiorino C, Dell'oca I, Broggi S, Cattaneo GM, Di Muzio N, Fazio F, Calandrino R, Schwarz M. Intensity-modulated proton therapy versus helical tomotherapy in nasopharynx cancer: planning comparison and NTCP evaluation. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):589-96. doi: 10.1016/j.ijrobp.2008.05.065. PMID 18793962
- [Background] Durante M, Loeffler JS. Charged particles in radiation oncology. Nat Rev Clin Oncol. 2010 Jan;7(1):37-43. doi: 10.1038/nrclinonc.2009.183. Epub 2009 Dec 1. PMID 19949433
- [Background] Moiseenko V, Wu J, Hovan A, Saleh Z, Apte A, Deasy JO, Harrow S, Rabuka C, Muggli A, Thompson A. Treatment planning constraints to avoid xerostomia in head-and-neck radiotherapy: an independent test of QUANTEC criteria using a prospectively collected dataset. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):1108-14. doi: 10.1016/j.ijrobp.2011.04.020. Epub 2011 Jun 2. PMID 21640505
- [Background] Beetz I, Schilstra C, van der Schaaf A, van den Heuvel ER, Doornaert P, van Luijk P, Vissink A, van der Laan BF, Leemans CR, Bijl HP, Christianen ME, Steenbakkers RJ, Langendijk JA. NTCP models for patient-rated xerostomia and sticky saliva after treatment with intensity modulated radiotherapy for head and neck cancer: the role of dosimetric and clinical factors. Radiother Oncol. 2012 Oct;105(1):101-6. doi: 10.1016/j.radonc.2012.03.004. Epub 2012 Apr 18. PMID 22516776
- [Background] Zhou X, Ou X, Xu T, Wang X, Shen C, Ding J, Hu C. Effect of dosimetric factors on occurrence and volume of temporal lobe necrosis following intensity modulated radiation therapy for nasopharyngeal carcinoma: a case-control study. Int J Radiat Oncol Biol Phys. 2014 Oct 1;90(2):261-9. doi: 10.1016/j.ijrobp.2014.05.036. Epub 2014 Jul 24. PMID 25066214
- [Background] Chan SH, Ng WT, Kam KL, Lee MC, Choi CW, Yau TK, Lee AW, Chow SK. Sensorineural hearing loss after treatment of nasopharyngeal carcinoma: a longitudinal analysis. Int J Radiat Oncol Biol Phys. 2009 Apr 1;73(5):1335-42. doi: 10.1016/j.ijrobp.2008.07.034. Epub 2008 Oct 14. PMID 18922648
- [Background] Wu LR, Liu YT, Jiang N, Fan YX, Wen J, Huang SF, Guo WJ, Bian XH, Wang FJ, Li F, Song D, Wu JF, Jiang XS, Liu JY, He X. Ten-year survival outcomes for patients with nasopharyngeal carcinoma receiving intensity-modulated radiotherapy: An analysis of 614 patients from a single center. Oral Oncol. 2017 Jun;69:26-32. doi: 10.1016/j.oraloncology.2017.03.015. Epub 2017 Apr 7. PMID 28559017
- [Background] Zheng Y, Han F, Xiao W, Xiang Y, Lu L, Deng X, Cui N, Zhao C. Analysis of late toxicity in nasopharyngeal carcinoma patients treated with intensity modulated radiation therapy. Radiat Oncol. 2015 Jan 13;10:17. doi: 10.1186/s13014-014-0326-z. PMID 25582731
- [Background] Tang LL, Guo R, Zhang N, Deng B, Chen L, Cheng ZB, Huang J, Hu WH, Huang SH, Luo WJ, Liang JH, Zheng YM, Zhang F, Mao YP, Li WF, Zhou GQ, Liu X, Chen YP, Xu C, Lin L, Liu Q, Du XJ, Zhang Y, Sun Y, Ma J. Effect of Radiotherapy Alone vs Radiotherapy With Concurrent Chemoradiotherapy on Survival Without Disease Relapse in Patients With Low-risk Nasopharyngeal Carcinoma: A Randomized Clinical Trial. JAMA. 2022 Aug 23;328(8):728-736. doi: 10.1001/jama.2022.13997. PMID 35997729
- [Background] Lv X, Cao X, Xia WX, Liu KY, Qiang MY, Guo L, Qian CN, Cao KJ, Mo HY, Li XM, Li ZH, Han F, He YX, Liu YM, Wu SX, Bai YR, Ke LR, Qiu WZ, Liang H, Liu GY, Miao JJ, Li WZ, Lv SH, Chen X, Zhao C, Xiang YQ, Guo X. Induction chemotherapy with lobaplatin and fluorouracil versus cisplatin and fluorouracil followed by chemoradiotherapy in patients with stage III-IVB nasopharyngeal carcinoma: an open-label, non-inferiority, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 May;22(5):716-726. doi: 10.1016/S1470-2045(21)00075-9. Epub 2021 Apr 12. PMID 33857411
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Kong L, Zhang Y, Hu C, Guo Y, Lu JJ. Effects of induction docetaxel, platinum, and fluorouracil chemotherapy in patients with stage III or IVA/B nasopharyngeal cancer treated with concurrent chemoradiation therapy: Final results of 2 parallel phase 2 clinical trials. Cancer. 2017 Jun 15;123(12):2258-2267. doi: 10.1002/cncr.30566. Epub 2017 Feb 13. PMID 28192641
- [Background] Tang LQ, Chen DP, Guo L, Mo HY, Huang Y, Guo SS, Qi B, Tang QN, Wang P, Li XY, Li JB, Liu Q, Gao YH, Xie FY, Liu LT, Li Y, Liu SL, Xie HJ, Liang YJ, Sun XS, Yan JJ, Wu YS, Luo DH, Huang PY, Xiang YQ, Sun R, Chen MY, Lv X, Wang L, Xia WX, Zhao C, Cao KJ, Qian CN, Guo X, Hong MH, Nie ZQ, Chen QY, Mai HQ. Concurrent chemoradiotherapy with nedaplatin versus cisplatin in stage II-IVB nasopharyngeal carcinoma: an open-label, non-inferiority, randomised phase 3 trial. Lancet Oncol. 2018 Apr;19(4):461-473. doi: 10.1016/S1470-2045(18)30104-9. Epub 2018 Feb 28. PMID 29501366
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945